CLINICAL TRIAL: NCT04399915
Title: Effect of Oxalate and Urate Metabolism on the Evolution of Kidney Disease
Brief Title: Effect of Oxalate and Urate Metabolism on CKD Evolution
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Institute of Nephrology of the Academy of Medical Sciences of Ukraine (Other)
Responsible Party: Sponsor
Other Study IDs: 0119U000002
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: CKD; ESRD; Hyperuricemia; Oxaluria
Keywords: CKD; hemodialysis; peritoneal dialysis; oxalate; uric acid; metabolism; renal survival; cardio-vascular events
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperuricemia; Hyperoxaluria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hyperoxalemia/Hyperuricemia Group
- Hyperoxalemia/Hyperuricemia-free Group
- Healthy Subjects

SUMMARY:
The current study primarily aimed to characterize the oxalate and uric acid metabolism in CKD patients and to analyze its association with renal survival prognosis. Secondarily, the study is planned to determine whether hyperoxalemia and hyperuricemia are independent risk factors for cardiovascular events and mortality.

DETAILED DESCRIPTION:
The study protocol is approved by a local Ethics Committee and registered in Domestic Clinical Trial Registry (Identifier 0119U000002). Writing informed consent is obtained from all subjects participating in the study.

The study will enroll 300 participants (250 CKD patients at stage 1-5 and 50 healthy subjects). Routine biochemical parameters including blood and daily dialysate concentration of urea and creatinine, serum albumin, C-reactive protein (CRP), glucose, electrolytes, and lipid profile parameters will carry out. Total oxalate-degrading activity in fecal samples, as well as plasma oxalic acid concentration, daily urinary oxalate excretion and peritoneal dialysis effluent oxalate concentration (if any) will determine. Uric acid will also measure in serum, urine and dialysate of peritoneal dialysis patients.

The study will be followed up for 3 years. The primary endpoint is cardiovascular events, secondary endpoints are dialysis adequacy and all-cause mortality. All the endpoints will be collected, as well as other outcomes, such as chronic inflammation, dyslipidemia and dialysis dose, and so on. The outcomes will be analyzed using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old,
* CKD stage 1-4,
* the patients did not take antibiotics and/or probiotics, lipid- and/or urate-lowering therapy for at least past 3 months or:
* dialysis treatment for at least 3 months,
* a stable clinical condition and adequately functioning arteriovenous fistula or peritoneal access,
* a target level of Kt/V (≥ 1.4 for the HD patients and ≥1.7 for the PD patients).

Exclusion Criteria:

* hospitalization in the preceding 3 months,
* previous history or actual diagnosis of peritonitis, anemia, systemic and malignant diseases, acute inflammation processes, immunosuppressive treatment and active hepatitis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD stage 1-5 patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Renal Survival for CKD stages 1-3 | 3 years

SECONDARY OUTCOMES:
Cardio-vascular Events | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Natalia Stepanova, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided